CLINICAL TRIAL: NCT04686058
Title: Propofol Patient-controlled Sedation Versus Target-controlled Infusion in Outpatient Colonoscopy
Brief Title: Sedation Techniques for Outpatient Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Nadia Md Nor, Primary Investigator, consultant anaesthesiologist, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FF-2014-203
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Colonoscopy
Keywords: TCI propofol; PCS propofol; sedation; colonoscopy
MeSH Terms: interventions — Propofol; Injections; Midazolam; Meperidine; Solutions

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TCI propofol (Active Comparator): Target controlled infusion propofol titrated by the investigator intra-procedure, based on the Modified Observer's Assessment of Alertness and Sedation Scale
  Interventions: Drug: Propofol 10 MG/ML Injection; Device: target controlled infusion pump
- PCS propofol (Active Comparator): Patient-controlled sedation titrated by the patient to comfort level
  Interventions: Drug: Propofol 10 MG/ML Injection; Device: patient-controlled sedation pump
- midazolam and pethidine (Active Comparator): Midazolam and pethidine bolus doses administered by the investigator based on clinical parameters and observation
  Interventions: Drug: Midazolam injection; Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection

INTERVENTIONS:
Drug: Propofol 10 MG/ML Injection
  Other Names: propofol
  Arms: PCS propofol; TCI propofol
Drug: Midazolam injection
  Other Names: midazolam
  Arms: midazolam and pethidine
Drug: Pethidine Hydrochloride 50 Mg/mL Solution for Injection
  Other Names: pethidine
  Arms: midazolam and pethidine
Device: target controlled infusion pump
  Other Names: TCI
  Arms: TCI propofol
Device: patient-controlled sedation pump
  Other Names: PCS
  Arms: PCS propofol

SUMMARY:
This was a prospective, randomized, single-blind controlled clinical trial comparing three sedative regimens for outpatient colonoscopy.

DETAILED DESCRIPTION:
This was a prospective, randomized, single-blind controlled clinical trial comparing target-controlled infusion (TCI) with propofol and patient-controlled sedation (PCS) with propofol, to conventional combination of midazolam and pethidine, in terms of quality and safety of sedation, and patient recovery during outpatient colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients
* aged between 18 to 80 years
* scheduled for outpatient colonoscopy

Exclusion Criteria:

* history of or with psychiatric disease
* on psychoactive drugs
* mentally or physically unable to use the hand-held device for PCS
* previous complications from anaesthesia or sedation
* potentially difficult airway maintenance
* obstructive sleep apnoea
* pregnant
* with contraindications to the study drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Recovery time to Modified Observer's Assessment of Alertness and Sedation Scale (MOAAS) | From time of arrival at the recovery area after completion of colonoscopy, until point of discharge from recovery area, assessed up to 2 hours post arrival at recovery
  Recovery of patient from sedation when MOAAS 5 is achieved
Recovery time to ambulation | From time of arrival at the recovery area after completion of colonoscopy, until the point patient starts to ambulate, assessed up to 2 hours post arrival at recovery
  Recovery of patient from sedation when patient starts ambulating
Recovery time to discharge | From time of arrival at the recovery area after completion of colonoscopy, until the point patient is deemed fit for discharge home, assessed up to 2 hours post arrival at recovery
  Recovery of patient from sedation when patient is deemed fit for discharge home
Endoscopist satisfaction score | After completion of colonoscopy, the endoscopist graded his satisfaction score from the start of colonoscopy, assessed until 2 hours after completion of colonoscopy
  After completion of colonoscopy, the endoscopist graded on a scale of 1 to 10, ease of the colonoscopy/procedure (1 = very difficult, 10 = very easy), and level of satisfaction (1 = very dissatisfied, 10 = very satisfied) using a 10 cm visual analog scale (VAS).
Patient satisfaction score | Patient satisfaction score from start of sedation until point of discharge from recovery assessed until 3 hours from the start of sedation
  After completion of colonoscopy, the patient graded on a scale of 1 to 10, the level of satisfaction (1 = very dissatisfied, 10 = very satisfied) using a 10 cm visual analog scale (VAS).
Patient willingness to repeat the same sedation technique | From patient arrival to recovery post colonoscopy, area until the point of patient discharge, assessed up to 3 hours after arrival at recovery
  Patient responds yes or no. to willingness of having the same sedation during colonoscopy, in the future

SECONDARY OUTCOMES:
Rescue analgesic drug requirement | From start of sedation, and during the entire duration of colonoscopy, assessed up to 2 hours from the start of sedation
  Requirement for rescue analgesic or sedative in addition to study drugs/sedatives, during the entire duration of colonoscopy
Total drug consumption | Total consumption of all study drugs from the start of sedation, during the entire duration of colonoscopy until completion of colonoscopy, assessed up to 2 hours from the start of sedation
  Total consumption of all study drugs from the start of sedation, during the entire duration of colonoscopy until completion of colonoscopy
Ease of colonoscopy score | during the entire duration of colonoscopy from the start of colonoscopy, assessed up to 2 hours from the start of colonoscopy
  endoscopist graded on a scale of 1 to 10, ease of procedure (1 = very difficult, 10 = very easy)
Recalled events during colonoscopy | Recalled events retrieved from patient, from arrival to recovery area until point of discharge home, assessed up to 2 hours from arrival at recovery
  The number of recalled events during the entire duration of colonoscopy
Recalled discomfort/ pain during colonoscopy | Recalled events of discomfort/pain retrived from the patient, from arrival to recovery area until point of discharge home, assessed up to 2 hours from arrival at recovery
  The number of recalled events of discomfor/pain during the entire duration of colonoscopy

OTHER OUTCOMES:
Time taken to onset of sedation | From start of sedation until MOAAS 3 or 4 attained, assessed up to one hour from the point sedation was commenced
  Time taken for patient to reach a sedation score of MOAAS 3 or 4

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No